CLINICAL TRIAL: NCT02781727
Title: A Multicenter, Phase 3, Randomized, Open-label, Active-controlled, Parallel-group Trial Investigating the Safety, Tolerability, and Efficacy of TransCon hGH Administered Once a Week Versus Standard Daily hGH Replacement Therapy Over 52 Weeks in Prepubertal Children With Growth Hormone Deficiency (GHD)
Brief Title: A Phase 3 Trial of the Safety, Tolerability and Efficacy of TransCon hGH Weekly Versus Daily hGH in Children With Growth Hormone Deficiency (GHD)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Ascendis Pharma Endocrinology Division A/S (Industry)
Responsible Party: Sponsor
Organization: Ascendis Pharma A/S (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TransCon hGH CT-301; 2016-001145-11 (EudraCT Number)
Record Dates: First submitted 2016-05-19; First posted 2016-05-24 (Estimated); Results first posted 2022-01-04 (Actual); Last update posted 2022-01-04 (Actual); Status verified 2021-12

CONDITIONS: Growth Hormone Deficiency, Pediatric; hGH (Human Growth Hormone); Endocrine System Diseases; Hormones; Pituitary Diseases
Keywords: Human Growth Hormone; hGH; GHD; rHGH; Pediatric Growth Hormone Deficiency; Long Acting Growth Hormone; Somatropin; Prodrug; Growth Failure; Growth Hormone Replacement Therapy; Sustained Release; Sustained Release Growth Hormone; Growth Hormone Deficiency
MeSH Terms: conditions — Dwarfism, Pituitary; Endocrine System Diseases; Pituitary Diseases; Failure to Thrive

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- TransCon hGH (Experimental): Once weekly subcutaneous injection of TransCon hGH
  Interventions: Drug: Once weekly subcutaneous injection of TransCon hGH
- human growth hormone (Genotropin) (Active Comparator): Once daily subcutaneous injection of Genotropin
  Interventions: Drug: Once daily subcutaneous injection of Genotropin

INTERVENTIONS:
Drug: Once weekly subcutaneous injection of TransCon hGH — Once weekly subcutaneous injection
  Arms: TransCon hGH
Drug: Once daily subcutaneous injection of Genotropin — Once daily subcutaneous injection
  Arms: human growth hormone (Genotropin)

SUMMARY:
A 52 week trial of TransCon hGH, a long-acting growth hormone product, versus human growth hormone therapy. TransCon hGH will be given once-a-week, human growth hormone (hGH) will be given daily. Approximately 150 prepubertal, hGH-treatment naïve children (males and females) with GHD will be included. Randomization will occur in a 2:1 ratio (TransCon hGH : Genotropin). This is a global trial that will be conducted in Armenia, Australia, Belarus, Bulgaria, Georgia, Greece, Italy, New Zealand, Poland, Romania, Russia, Turkey, Ukraine, and the United States.

ELIGIBILITY:
Inclusion Criteria:

* Prepubertal children with GHD (either isolated or as part of a multiple pituitary hormone deficiency) in Tanner stage 1 (Tanner 1982) aged:

  * Boys: 3-12 years, inclusive
  * Girls: 3-11 years, inclusive
* Impaired height (HT) defined as at least 2.0 standard deviations (SD) below the mean height for chronological age and sex (HT SDS ≤ -2.0) according to the 2000 CDC Growth Charts for the United States Methods and Development, available at http://www.cdc.gov/growthcharts/
* Diagnosis of GHD confirmed by 2 different GH stimulation tests, defined as a peak GH level of ≤10 ng/mL, determined with a validated assay
* Bone age (BA) at least 6 months less than chronological age
* Baseline IGF-1 level of at least 1 SD below the mean IGF-1 level standardized for age and sex (IGF-1 SDS ≤-1)
* Written, signed informed consent of the parent(s) or legal guardian(s) of the subject and written assent of the subject (if the subject is able to read, understand, and sign)

Exclusion Criteria:

* Children with a body weight below 12 kg
* Prior exposure to recombinant hGH or IGF-1 therapy
* Children with past or present intracranial tumor growth as confirmed by a sellar MRI scan (with contrast) at Screening (MRI results from up to 6 months prior to Screening may be accepted)
* Children with psychosocial dwarfism
* Children with idiopathic short stature
* History or presence of malignant disease; any evidence of present tumor growth
* Closed epiphyses
* Major medical conditions and/or presence of contraindication to hGH treatment
* Participation in any other trial of an investigational agent within 3 months prior to Screening

Ages: 3 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 162 (Actual)
Dates: Start 2016-12-13 (Actual); Primary Completion 2019-01-17 (Actual); Study Completion 2019-01-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Beckert, MD, Study Director — Ascendis Pharma A/S; Aimee D Shu, MD, Study Director — Ascendis Pharma, Inc.
Locations (48):
- United States (16):
  - Ascendis Pharma Investigational Site, Birmingham, Alabama
  - Ascendis Pharma Investigational Site, Little Rock, Arkansas
  - Ascendis Pharma Investigational Site, Los Angeles, California
  - Ascendis Pharma Investigational Site, Orange, California
  - Ascendis Pharma Investigational Site, Centennial, Colorado
  - Ascendis Pharma Investigational Site, Jacksonville, Florida
  - Ascendis Pharma Investigational Site, Orlando, Florida
  - Ascendis Pharma Investigational Site, Saint Paul, Minnesota
  - Ascendis Pharma Investigational Site, Jackson, Mississippi
  - Ascendis Pharma Investigational Site, Lebanon, New Hampshire
  - Ascendis Pharma Investigational Site, Mineola, New York
  - Ascendis Pharma Investigational Site, Oklahoma City, Oklahoma
  - Ascendis Pharma Investigational Site, Portland, Oregon
  - Ascendis Pharma Investigational Site, Dallas, Texas
  - Ascendis Pharma Investigational Site, Fort Worth, Texas
  - Ascendis Pharma Investigational Site, Tacoma, Washington
- Ascendis Pharma Investigational Site, Yerevan, Armenia
- Ascendis Pharma Investigational Site, Clayton, Australia
- Ascendis Pharma Investigational Site, Minsk, Belarus
- Ascendis Pharma Investigational Site, Varna, Bulgaria
- Ascendis Pharma Investigational Site, Tbilisi, Georgia
- Ascendis Pharma Investigational Site, Athens, Greece
- Italy (2):
  - Ascendis Pharma Investigational Site, Milan
  - Ascendis Pharma Investigational Site, Roma
- Ascendis Pharma Investigational Site, Grafton, New Zealand
- Poland (2):
  - Ascendis Pharma Investigatonal Site, Gdansk
  - Ascendis Pharma Investigational Site, Warsaw
- Ascendis Pharma Investigational Site, Iași, Romania
- Russia (14):
  - Ascendis Pharma Investigational Site, Izhevsk
  - Ascendis Pharma Investigational Site, Kazan'
  - Ascendis Pharma Investigational Site, Krasnoyarsk
  - Ascendis Pharma Investigational Site, Moscow
  - Ascendis Pharma Investigational Site, Nizhny Novgorod
  - Ascendis Pharma Investigational Site, Novosibirsk
  - Ascendis Pharma Investigational Site, Omsk
  - Ascendis Pharma Investigational Site, Saint Petersburg
  - Ascendis Pharma Investigational Site, Samara
  - Ascendis Pharma Investigational Site, Saratov
  - Ascendis Pharma Investigational Site, Tomsk
  - Ascendis Pharma Investigational Site, Ufa
  - Ascendis Pharma Investigational Site, Vologda
  - Ascendis Pharma Investigational Site, Voronezh
- Turkey (Türkiye) (3):
  - Ascendis Pharma Investigational Site, Izmir
  - Ascendis Pharma Investigational Site, Melikgazi
  - Ascendis Pharma Investigational Site, Trabzon
- Ukraine (3):
  - Ascendis Pharma Investigational Site, Kharkiv
  - Ascendis Pharma Investigational Site, Kyiv
  - Ascendis Pharma Investigational Site, Odesa

REFERENCES:
- [Derived] Thornton PS, Maniatis AK, Aghajanova E, Chertok E, Vlachopapadopoulou E, Lin Z, Song W, Christoffersen ED, Breinholt VM, Kovalenko T, Giorgadze E, Korpal-Szczyrska M, Hofman PL, Karpf DB, Shu AD, Beckert M. Weekly Lonapegsomatropin in Treatment-Naive Children With Growth Hormone Deficiency: The Phase 3 heiGHt Trial. J Clin Endocrinol Metab. 2021 Oct 21;106(11):3184-3195. doi: 10.1210/clinem/dgab529. PMID 34272849

RESULTS

PARTICIPANT FLOW:
Groups:
- Lonapegsomatropin: Once weekly subcutaneous injection of lonapegsomatropin (TransCon hGH)
- Daily hGH: Once daily subcutaneous injection of Genotropin
Period: Pre-dosing Period
Arm/Group | Lonapegsomatropin | Daily hGH
Started | 106 (106 subjects were randomized to the lonapegsomatropin arm, but 1 subject withdrew consent before receiving the first dose of study drug.) | 56
Completed | 105 | 56
Not Completed | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0
Period: Treatment Period
Arm/Group | Lonapegsomatropin | Daily hGH
Started | 105 | 56
Completed | 104 | 55
Not Completed | 1 | 1
Not completed — Withdrawal by Subject | 1 | 0
Not completed — Lost to Follow-up | 0 | 1

BASELINE CHARACTERISTICS:
Population: The Intention-to-Treat (ITT) population included all randomized subjects who had received at least 1 dose of active treatment.
Groups:
- Total: Total of all reporting groups
Arm/Group | Lonapegsomatropin | Daily hGH | Total
Number analyzed (Participants) | 105 | 56 | 161
Age, Continuous [Mean (Standard Deviation); unit: years] | 8.5 (2.7) | 8.5 (2.8) | 8.5 (2.7)
Age, Customized [Count of Participants; unit: Participants]
  Age, Categorical: <6 years | 25 | 14 | 39
  Age, Categorical: ≥6 years | 80 | 42 | 122
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19 | 10 | 29
  Male | 86 | 46 | 132
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: Asian | 1 | 0 | 1
  Race: Black or African American | 2 | 1 | 3
  Race: White | 100 | 52 | 152
  Race: Other | 2 | 3 | 5
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Ethnicity: Hispanic or Latino | 5 | 2 | 7
  Ethnicity: Not Hispanic or Latino | 100 | 54 | 154
Height [Mean (Standard Deviation); unit: cm] | 112.93 (14.09) | 112.15 (15.29) | 112.66 (14.48)
Height SDS [Mean (Standard Deviation); unit: standard deviation score] — Height Standard Deviation Score (SDS) is the number of standard deviations above or below the mean height for age and sex. Height SDS was derived using the LMS method as ((Height/M)^L)-1)/(L x S), where M = median, S = generalized coefficient of variation, and L = power in the Box-Cox transformation, the M, S, L values were obtained from 2000 CDC growth charts for the United States. A Standard Deviation Score of 0 represents the population mean.
  standard deviation score | -2.89 (0.85) | -3.00 (0.90) | -2.93 (0.87)
Weight [Mean (Standard Deviation); unit: kg] | 21.01 (6.54) | 21.20 (6.67) | 21.08 (6.56)
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] | 16.06 (1.78) | 16.46 (2.17) | 16.20 (1.93)
BMI SDS [Mean (Standard Deviation); unit: standard deviation score] — BMI Standard Deviation Score (SDS) is the number of standard deviations above or below the mean body mass index for age and sex. BMI SDS was derived using the LMS method as ((BMI/M)^L)-1)/(L x S), where M = median, S = generalized coefficient of variation, and L = power in the Box-Cox transformation, the M, S, L values were obtained from 2000 CDC growth charts for the United States. A Standard Deviation Score of 0 represents the population mean.
  standard deviation score | -0.32 (0.95) | -0.14 (1.07) | -0.25 (0.99)
IGF-1 SDS [Mean (Standard Deviation); unit: standard deviation score] — IGF-1 Standard Deviation Score (SDS) is the number of standard deviations above or below the mean Insulin-like Growth Factor 1 (IGF-1) level for age and sex. IGF-1 SDS was derived using the LMS method as ((IGF-1/M)^L)-1)/(L x S), where M = median, S = generalized coefficient of variation, and L = power in the Box-Cox transformation, the M, S, L values were obtained from Bidlingmaier et al. (2014). A Standard Deviation Score of 0 represents the population mean.
  standard deviation score | -2.08 (0.88) | -1.96 (0.98) | -2.04 (0.92)

OUTCOME MEASURES:

1. Primary Outcome: Annualized Height Velocity at 52 Weeks for Weekly Lonapegsomatropin and Daily hGH Treatment Groups
Description: Annualized height velocity (AHV) at 52 weeks for weekly lonapegsomatropin (TransCon hGH) and daily hGH treatment groups
Time Frame: 52 weeks
Population: as for baseline characteristics
Measure: Least Squares Mean (Standard Error); unit: cm/year
Arm/Group | Lonapegsomatropin | Daily hGH
Number analyzed (Participants) | 105 | 56
cm/year | 11.17 (0.23) | 10.31 (0.30)
Statistical Analysis 1: Comparison: Lonapegsomatropin vs Daily hGH; ANCOVA model with multiple imputation. For each imputed data set, an ANCOVA model with by visit AHV as the dependent variable; treatment and gender as factors; and baseline age, baseline peak GH levels (log transformed) at stimulation test, and baseline height SDS - average parental height SDS as covariates were fitted; Test type: Non-Inferiority — Non-inferiority comparison with a non-inferiority margin of 2 cm/year, followed by a test of superiority if non-inferiority is established; p = 0.0088, ANCOVA with multiple imputation — P-value is based on a test of superiority; two-sided

2. Secondary Outcome: Number of Participants With Treatment-Emergent Adverse Events [Safety and Tolerability]
Description: Number of participants with Treatment-Emergent Adverse Events for the weekly lonapegsomatropin and daily hGH treatment groups
Time Frame: 52 Weeks
Population: The safety analysis population included all randomized subjects who had received at least 1 dose of active treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Lonapegsomatropin | Daily hGH
Number analyzed (Participants) | 105 | 56
Participants
  TEAEs | 81 | 39
  TEAEs related to study drug | 12 | 10
  SAEs | 1 | 1
  SAEs related to study drug | 0 | 0

3. Secondary Outcome: Annualized Height Velocity Over 52 Weeks for Weekly Lonapegsomatropin and Daily hGH Treatment Groups
Description: Annualized height velocity (AHV) over 52 weeks for weekly lonapegsomatropin and daily hGH treatment groups. AHV by visit was determined by ANCOVA model with multiple imputation. For each imputed data set, an ANCOVA model with by visit AHV as the dependent variable, treatment and gender as factors, baseline age, baseline peak GH levels (log transformed) at stimulation test, and baseline height SDS - average parental height SDS as covariates were fitted.
Time Frame: Week 5, Week 13, Week 26, Week 39 and Week 52
Population: as for baseline characteristics
Measure: Least Squares Mean (Standard Error); unit: cm/year
Arm/Group | Lonapegsomatropin | Daily hGH
Number analyzed (Participants) | 105 | 56
cm/year
  Week 5 | 13.54 (1.07) | 12.83 (1.37)
  Week 13 | 13.28 (0.49) | 12.22 (0.63)
  Week 26 | 12.65 (0.32) | 11.21 (0.42)
  Week 39 | 11.89 (0.26) | 10.90 (0.33)
  Week 52 | 11.17 (0.23) | 10.31 (0.30)

4. Secondary Outcome: Change in Height Standard Deviation Score Over 52 Weeks for the Weekly Lonapegsomatropin and Daily hGH Treatment Groups
Description: Height Standard Deviation Score (SDS) is the number of standard deviations above or below the mean height for age and sex. Height SDS was derived using the LMS method as ((Height/M)^L)-1)/(L x S), where M = median, S = generalized coefficient of variation, and L = power in the Box-Cox transformation, the M, S, L values were obtained from 2000 CDC growth charts for the United States. A Standard Deviation Score of 0 represents the population mean. A higher change from baseline in Height Standard Deviation Score (SDS) indicates a better outcome. The change from baseline in height SDS by visit was determined by ANCOVA model and included baseline age, peak GH levels (log transformed) at stimulation test and baseline height SDS as covariates, as well as treatment and gender as factors.
Time Frame: Week 5, Week 13, Week 26, Week 39 and Week 52
Population: as for baseline characteristics
Measure: Least Squares Mean (Standard Error); unit: standard deviation score
Arm/Group | Lonapegsomatropin | Daily hGH
Number analyzed (Participants) | 105 | 56
standard deviation score
  Week 5 | 0.13 (0.02) | 0.12 (0.02)
  Week 13 | 0.38 (0.02) | 0.33 (0.03)
  Week 26 | 0.68 (0.03) | 0.58 (0.04)
  Week 39 | 0.92 (0.03) | 0.80 (0.04)
  Week 52 | 1.10 (0.04) | 0.96 (0.05)

5. Secondary Outcome: Average IGF-1 Standard Deviation Score Over 52 Weeks for the Weekly Lonapegsomatropin and Daily hGH Treatment Groups
Description: IGF-1 Standard Deviation Score (SDS) is the number of standard deviations above or below the mean Insulin-like Growth Factor 1 (IGF-1) level for age and sex. IGF-1 SDS was derived using the LMS method as ((IGF-1/M)^L)-1)/(L x S), where M = median, S = generalized coefficient of variation, and L = power in the Box-Cox transformation, the M, S, L values were obtained from Bidlingmaier et al. (2014). A Standard Deviation Score of 0 represents the population mean. Average IGF-1 SDS by visit was determined by ANCOVA. The ANCOVA model included baseline age, peak GH levels (log transformed) at stimulation test, baseline IGF-1 SDS as covariates, as well as treatment and gender as factors. Modeled values begin at Week 13 corresponding with achievement of IGF-1 steady state. Average IGF-1 SDS values by visit for the Lonapegsomatropin group were derived from a population pharmacodynamic model; the average IGF-1 SDS values for the Genotropin group are represented by observed values.
Time Frame: Week 13, Week 26, Week 39, and Week 52
Population: as for baseline characteristics
Measure: Least Squares Mean (Standard Error); unit: standard deviation score
Arm/Group | Lonapegsomatropin | Daily hGH
Number analyzed (Participants) | 105 | 56
standard deviation score
  Week 13 | 0.31 (0.09) | -0.60 (0.11)
  Week 26 | 0.46 (0.08) | -0.51 (0.10)
  Week 39 | 0.59 (0.09) | -0.30 (0.11)
  Week 52 | 0.72 (0.09) | -0.02 (0.12)

6. Secondary Outcome: Number of Participants With Treatment Emergent Anti-hGH Binding Antibody Formation
Description: Number of participants with treatment emergent anti-hGH binding antibody formation during the 52 week study. All samples were negative for anti-hGH neutralizing antibodies.
Time Frame: Start of study treatment through Week 52
Population: The safety analysis population included all randomized subjects who had received at least 1 dose of active treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Lonapegsomatropin | Daily hGH
Number analyzed (Participants) | 105 | 56
Participants | 6 | 2

ADVERSE EVENTS:
Time Frame: From the first trial-related activity after the subject signed the informed consent until the end of the post-treatment follow-up period (up to week 52)
Description: All adverse events (AEs) were collected in response to a general question about the subject's well-being and any possible changes from the previous visit, but were not specifically solicited. AEs, including any serious adverse events, were collected through the end of trial (ie, the Week 52 Visit 6). AEs ongoing at Visit 6 or the time of premature trial discontinuation were followed until the event was resolved or deemed stable by the investigator.
Arm/Group | Lonapegsomatropin | Daily hGH
All-Cause Mortality (participants affected / at risk) | 0/105 | 0/56
Serious Adverse Events (participants affected / at risk) | 1/105 | 1/56
Other Adverse Events (participants affected / at risk) | 81/105 | 39/56
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Lonapegsomatropin (N=105) | Daily hGH (N=56)
Appendicitis (Infections and infestations) | 1 | 0
Concussion (Injury, poisoning and procedural complications) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Lonapegsomatropin (N=105) | Daily hGH (N=56)
Nasopharyngitis (Infections and infestations) | 12 | 8
Pharyngitis (Infections and infestations) | 10 | 10
Upper respiratory tract infection (Infections and infestations) | 6 | 5
Respiratory tract infection (Infections and infestations) | 7 | 3
Cough (Respiratory, thoracic and mediastinal disorders) | 10 | 4
Vomiting (Gastrointestinal disorders) | 9 | 3
Diarrhea (Gastrointestinal disorders) | 6 | 3
Pyrexia (General disorders) | 16 | 5
Headache (Nervous system disorders) | 13 | 7
Secondary hypothyroidism (Endocrine disorders) | 7 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2017-09-12): https://cdn.clinicaltrials.gov/large-docs/27/NCT02781727/Prot_000.pdf
  • Statistical Analysis Plan (2019-02-19): https://cdn.clinicaltrials.gov/large-docs/27/NCT02781727/SAP_001.pdf